CLINICAL TRIAL: NCT06959927
Title: Risk Factors and Application of Risk Management Strategies in Hemodialysis Patients Complicated With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guiren Hou (Other Government)
Responsible Party: Sponsor-Investigator, Guiren Hou, Principal Investigator, Changsha Fourth Hospital
Organization: Changsha Fourth Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: No. DSYY-2024-26
Record Dates: First submitted 2025-03-27; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Hemodialysis; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care Group (Other): Patients in this group received conventional hemodialysis care, including:
  Continuous monitoring of vital signs (blood pressure, respiratory rate, pulse, heart rhythm); Supplemental oxygen therapy as needed; Instruction on effective coughing techniques; Strict fluid and electrolyte management; Metabolic support therapies; Positional adjustments (upright posture with lower limb dependency); Environmental regulation (temperature: 22-24°C; humidity: 50-60%); Individualized dietary counseling.
  Interventions: Other: Standard Care Group
- Risk-Stratified Management Group (Other): Patients in this group received standard care plus targeted risk management interventions:
  System Enhancement:
  Standardized nursing protocols and accountability frameworks Competency-based staff training (emergency response, fluid management) Individualized care plans (e.g., intensified glycemic control for diabetics, optimized BP monitoring for hypertensives)
  Risk Stratification:
  Admission assessments and follow-up evaluations to identify high-risk patients Hemodynamic monitoring with alert thresholds for early deterioration detection Strict pharmacological supervision and fluid balance protocols
  Environmental Modification:
  Optimized dialysis unit conditions (temperature: 22-24°C; humidity: 50-60%) Dedicated cardiac care zones for HF patients
  Quality Control:
  Quarterly audits of critical care domains (patient education, vital signs documentation, protocol compliance, satisfaction metrics) Corrective actions for identified deficiencies
  Interventions: Other: Risk-Stratified Management Group

INTERVENTIONS:
Other: Standard Care Group — Patients in this group received conventional hemodialysis care, including:
  Continuous monitoring of vital signs (blood pressure, respiratory rate, pulse, heart rhythm); Supplemental oxygen therapy as needed; Instruction on effective coughing techniques; Strict fluid and electrolyte management; Metabolic support therapies; Positional adjustments (upright posture with lower limb dependency); Environmental regulation (temperature: 22-24°C; humidity: 50-60%); Individualized dietary counseling.
  Arms: Standard Care Group
Other: Risk-Stratified Management Group — Patients in this group received standard care plus targeted risk management interventions:
  System Enhancement:
  Standardized nursing protocols and accountability frameworks Competency-based staff training (emergency response, fluid management) Individualized care plans (e.g., intensified glycemic control for diabetics, optimized BP monitoring for hypertensives)
  Risk Stratification:
  Admission assessments and follow-up evaluations to identify high-risk patients Hemodynamic monitoring with alert thresholds for early deterioration detection Strict pharmacological supervision and fluid balance protocols
  Environmental Modification:
  Optimized dialysis unit conditions (temperature: 22-24°C; humidity: 50-60%) Dedicated cardiac care zones for HF patients
  Quality Control:
  Quarterly audits of critical care domains (patient education, vital signs documentation, protocol compliance, satisfaction metrics) Corrective actions for identified deficiencies
  Arms: Risk-Stratified Management Group

SUMMARY:
Age, hyperglycemia, inflammation, and comorbidities (hypertension, diabetes, coronary disease) independently increase HF risk in hemodialysis patients. Targeted risk management reduces psychological distress, complications, and enhances care outcomes.

DETAILED DESCRIPTION:
To identify risk factors for heart failure (HF) in hemodialysis patients and assess the efficacy of targeted risk management strategies in improving prognosis and care quality. A total of 170 hospitalized dialysis patients from January 2022 to January 2024 were enrolled. They were divided into two groups based on the presence or absence of heart failure: the heart failure group (n=80) and the non-heart failure group (n=90). The inducing factors were analyzed, and targeted risk management strategies were implemented, with the participants further divided into a conventional group (n=40) and a study group (n=40) to explore the effect of these strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients were aged 18 years or older who had been undergoing regular hemodialysis treatment for more than three months.

  * Patients were in good cardiopulmonary health without severe acute or chronic diseases, and were capable of undergoing the study-related examinations and treatments.

    * Patients had not undergone major surgeries or experienced acute complications within the three months prior to enrollment, and their conditions were stable.

      * Patients demonstrated high compliance by following medical advice and regularly attending dialysis sessions and related examinations.

        ⑤Patients were able to understand the study objectives, had signed the informed consent form, and were willing to cooperate with follow-up visits and long-term observation.

Exclusion Criteria:

* Patients were excluded if they had severe liver diseases (e.g., cirrhosis or liver failure), significant systemic infections, active tuberculosis, malignant tumors, connective tissue diseases, or other major illnesses.

  * Patients with congenital kidney diseases, congenital heart defects, or other severe congenital structural abnormalities were excluded.

    * Patients who had a documented history of severe cardiac diseases were excluded, including those with primary/secondary cardiomyopathy, valvular heart disease, myocarditis, or pericardial diseases.

      * Patients were excluded if they had severe mental disorders or cognitive impairments that prevented their cooperation with study assessments or treatments.

        ⑤Patients whose clinical records or examination data were incomplete, thereby precluding effective analysis, were excluded.

Ages: 38 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiac Events (MACE) in Hemodialysis Patients with Heart Failure | From enrollment until first occurrence of any MACE component, assessed over 12 months.
  Composite endpoint including:
  Cardiovascular mortality (death due to heart failure, myocardial infarction, or arrhythmia).
  Hospitalization for worsening heart failure (requiring IV diuretics, vasodilators, or mechanical support).
  Dialysis-related cardiovascular complications (e.g., intradialytic hypotension, arrhythmias).

SECONDARY OUTCOMES:
Change in Inflammatory Biomarkers | Baseline, 3 months, and 6 months.
  Reduction in serum C-reactive protein (CRP) and interleukin-6 (IL-6) levels from baseline to 6 months.
Glycemic Control Improvement | Baseline and 6 months.
  Absolute change in glycated hemoglobin (HbA1c) levels in diabetic patients.
Change in Psychological Distress (SAS/SDS Scores) | Baseline, 6, 12, and 24 months
  Reduction in anxiety/depression scores post-intervention:
  Self-rating Anxiety Scale (SAS; range 0-100, higher = worse)
  Self-rating Depression Scale (SDS; range 0-100, higher = worse)
Complication Rates | Over 12 months.
  Incidence of dialysis-related complications (hypotension, pulmonary edema, infections).
Nursing Satisfaction Score | 24 months
  Patient-reported satisfaction (25-item Likert scale; 1-4 per item, total 25-100; higher = better), categorized as:
  Very satisfied (>90)
  Satisfied (70-90)
  Dissatisfied (<70)

OTHER OUTCOMES:
Biomarker Correlates (HbA1c, CRP) | Baseline, 12, and 24 months
  Association between baseline HbA1c (>5.7%)/CRP (>3 mg/L) and HF incidence.
Hospitalization Frequency | 24 months
  All-cause and HF-related hospital admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Guiren Hou, MB, Principal Investigator — Changsha Fourth Hospital
Locations (1):
- Changsha Fourth Hospital, Changsha, China

IPD SHARING:
Plan to Share IPD: No